CLINICAL TRIAL: NCT02361476
Title: Does Intraoperative Clonidine Reduce Post Operative Agitation in Children Anaesthetised With Sevoflurane? A RCT Including Pharmacokinetic Investigation.
Brief Title: Does Intraoperative Clonidine Reduce Post Operative Agitation in Children?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mogens Ydemann, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H - 2 - 2014 - 072
Record Dates: First submitted 2015-02-01; First posted 2015-02-11 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-09

CONDITIONS: Psychomotor Agitation
Keywords: Anaesthesia; Children; Clonidine; Sevoflurane; Postoperative agitation; Prevention; Pharmacokinetics; Safety
MeSH Terms: conditions — Psychomotor Agitation | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Clonidine : injection og 3 micg/kg IV during the operation.
  Interventions: Drug: Clonidine
- Placebo (Placebo Comparator): Placebo : injection og equal amount of NaCl IV during the operation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine — Injection - during surgery
  Other Names: catapresan
  Arms: Intervention
Drug: Placebo — Injection - during surgery
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
Clonidine is widely used off-label in children for several indications. Clonidine is used for treatment and/or prevention of postoperative agitation in children anaesthetised with Sevoflurane. The investigators don´t have solid evidence for the effect and the investigators don´t have data for characterization of the pharmacokinetic profile among age-groups for children 1-6 years.

In this study the investigators want to investigate if IV Clonidine administered at the end of surgery can prevent/reduce postoperative agitation. Secondary outcomes include measurements of postoperative pain relief and adverse effects, including a 30-day follow-up.

DETAILED DESCRIPTION:
BACKGROUND:

Clonidine is widely used off-label in children for several indications such as treatment and/or prevention of postoperative agitation when anaesthetised with Sevoflurane. However, the current level of evidence in support of Clonidine treatment for postoperative agitation in children remains limited. In addition, the pharmacokinetic profile of intravenous Clonidine in children is not well characterized for age-groups.

METHODS/DESIGN:

In this prospective multicentre double-blinded randomized clinical trial, the investigators aim to investigate the impact of intravenous (IV) Clonidine administered at the end of surgery, on the incidence and degree of postoperative agitation. Children will be assigned to either the intervention or the placebo group. The allocation will be carried out centrally and stratified based on age and trial-site, with152 patients allocated to each group. In the intervention group, 3 micrograms per kg of IV clonidine is administered approximately 20 minutes before the expected completion of the surgery (as assessed by the surgeon). In the control group; Saline (placebo) is injected in equal quantity during surgery at the same time. The drugs are concealed in identical blinded ampoules.

The primary outcome is postoperative agitation measured on the Watcha scale. Secondary outcomes include measurements of postoperative pain relief and adverse effects, including 30-day follow-up.

Twenty of the patients age 1-2 years and twenty age >2 years, with a peripheral venous access in place, will be allocated to drug assay sampling; enabling a compartmental PK analysis based on age group, using non-linear mixed effects models.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for surgery with Sevoflurane as the choice of anesthesia.

Exclusion Criteria:

* ASA classification >2
* Premedication with Clonidine
* Ex-premature (born before week 37+0 AND <60 weeks old)
* Intubated before anaesthesia and/or no plans for extubation after anaesthesia.
* Critical illness with haemodynamic instability.
* Active bleeding.
* Cancer.
* Cardiac diseases including arrhythmias.
* Malignant hyperthermia.
* Mental retardation.
* Neurological illness with agitation-like symptoms.
* Weight >50 kg.
* Allergy to Clonidine.
* Patients treated with methylphenidate / Concerta.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 379 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steen Henneberg, MD, DMSc, Study Director — Rigshospitalet, Denmark
Locations (3):
- Denmark (3):
  - The Juliane Marie Centre, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Region Sjælland
  - Køge Sygehus, Anæstesiologisk Afdeling, Køge
  - Anæstesiologisk afdeling, Vejle Sygehus, Vejle

REFERENCES:
- [Background] Pickard A, Davies P, Birnie K, Beringer R. Systematic review and meta-analysis of the effect of intraoperative alpha(2)-adrenergic agonists on postoperative behaviour in children. Br J Anaesth. 2014 Jun;112(6):982-90. doi: 10.1093/bja/aeu093. Epub 2014 Apr 11. PMID 24727829
- [Derived] Ydemann M, Nielsen BN, Henneberg S, Jakobsen JC, Wetterslev J, Lauritsen T, Steen N, Edstrom B, Afshari A; PREVENT AGITATION Research Group. Intraoperative clonidine for prevention of postoperative agitation in children anaesthetised with sevoflurane (PREVENT AGITATION): a randomised, placebo-controlled, double-blind trial. Lancet Child Adolesc Health. 2018 Jan;2(1):15-24. doi: 10.1016/S2352-4642(17)30127-X. Epub 2017 Nov 2. PMID 30169192
- [Derived] Ydemann M, Nielsen BN, Wetterslev J, Henneberg S, Lauritsen T, Steen N, Edstrom B, Afshari A. Effect of clonidine to prevent agitation in children after sevoflurane anaesthesia: a randomised placebo controlled multicentre trial. Dan Med J. 2016 Jun;63(6):A5234. PMID 27264945

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Placebo
Started | 191 | 188
Completed | 191 | 188
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 191 | 188 | 379
Age, Customized [Number; unit: participants]
  < 2 years | 46 | 43 | 89
  >/= 2 years | 145 | 145 | 290
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 154 | 150 | 304
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 191 | 188 | 379

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Agitation
Description: Measured by Watchae Scale (score 1-4), scores 1-2 = no agitation and scores 3-4 = agitated
Time Frame: 1 day
Population: 9 were excluded in the primary outcome due to missing data points
Measure: Number; unit: participants with agitation
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 187 | 183
participants with agitation | 46 | 86

2. Secondary Outcome: Fentanyl and Morphine Requirements
Description: Amount used
Time Frame: Recorded during the stay in the postoperative recovery room
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 191 | 188
mg morphine equivalents | 0.46 (0.94) | 0.7 (1.11)

3. Secondary Outcome: Pain Assessment
Description: Pain score used:
  FLACC score = Face, Legs, Activity, Cry, Consolability Score ranges from 0 to 10 (severity increases with increasing score) Pain is FLACC score more than 3
Time Frame: recovery room - hours
Measure: Mean (Standard Deviation); unit: Pain Score
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 191 | 188
Pain Score | 1.57 (2.62) | 2.45 (3.1)

4. Secondary Outcome: First Administration of Fentanyl or Morphine
Description: Time to administration
Time Frame: recovery room
Measure: Median (Standard Deviation); unit: MEDIAN time (min) to administration
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 191 | 188
MEDIAN time (min) to administration | 105 (57) | 60 (46)

5. Secondary Outcome: Adverse Events
Time Frame: from intervention to discharge from the recovery room
Measure: Number; unit: participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 191 | 188
participants
  adverse events | 0 | 5
  serious adverse events | 2 | 2
  Treated for low blood pressure | 0 | 0

ADVERSE EVENTS:
Arm/Group | Intervention | Placebo
All-Cause Mortality (participants affected / at risk) | 0/191 | 0/188
Serious Adverse Events (participants affected / at risk) | 2/191 | 2/188
Other Adverse Events (participants affected / at risk) | 0/191 | 5/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=191) | Placebo (N=188)
Re-bleeding (Surgical and medical procedures) | 0 (0) | 1 (1) — events leading to admission
Late arrival in the postoperative care unit (General disorders) | 0 (0) | 1 (1) — events leading to admission
Pale and not drinking and eating (General disorders) | 1 (1) | 0 (0) — events leading to admission
PONV (Gastrointestinal disorders) | 1 (1) | 0 (0) — events leading to admission
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=191) | Placebo (N=188)
Opioid-related side-effects (General disorders) | 0 (0) | 3 (3)
Laryngeal spasm (General disorders) | 0 (0) | 1 (1)
Prolonged anaesthesia (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No